CLINICAL TRIAL: NCT01185600
Title: Microparticles in Stored Red Blood Cells (RBC) as Potential Mediators of Transfusion Complications (II): Clinical Study
Brief Title: Microparticles in Stored RBC as Potential Mediators of Transfusion Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Wenche Jy, Research Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20090685; R01HL098031 (NIH)
Record Dates: First submitted 2010-08-17; First posted 2010-08-20 (Estimated); Results first posted 2016-11-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Coronary Artery Bypass
Keywords: transfusion complications; washed RBC; microparticles; storage lesion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transfusion with washed RBC (Active Comparator): Subject assigned to this arm will be transfused with washed RBC
  Interventions: Biological: Washed RBC
- Transfusion with unwashed RBC (Active Comparator): Subjects assigned to this arm will be transfused with unwashed RBC
  Interventions: Biological: Unwashed RBC

INTERVENTIONS:
Biological: Washed RBC — There is no pre-set dosage, frequency and duration for transfusion with washed RBC. It all depends on the conditions of patients during and after surgery. As circumstances arise, the physician will request needed washed RBC for the subject.
  Other Names: Washed packed cells
  Arms: Transfusion with washed RBC
Biological: Unwashed RBC — There is no pre-set dosage, frequency and duration for transfusion with unwashed RBC. It all depends on the conditions of patients during and after surgery. As circumstances arise, the physician will request needed unwashed RBC for the subject.
  Other Names: Unwashed packed cells
  Arms: Transfusion with unwashed RBC

SUMMARY:
INTRODUCTION. Cell-derived microparticles (MP) are released in cell activation, apoptosis and other processes. MP derived from red cells (RMP) are known to be released from stored packed red blood cells (PRBC), and their number increases with storage time. This constitutes one aspect of the storage lesion. Adverse transfusion events are known to increase with time of PRBC storage. The explanation for this is not known.

HYPOTHESIS. Based on their findings and those of others, the investigators propose to test the hypothesis that MP in stored PRBC contribute to adverse effects of transfusion. Specifically, MP in stored blood: (1) increase procoagulant activity, expression of pro-inflammatory mediators, immune suppression, and endothelial disturbance; and (2) increase the risk of transfusion and post-operative complications in patients undergoing coronary artery bypass grafting (CABG).

AIMS & PROCEDURES. The aim of this study is to assess the clinical significance of MPs in PRBC-related transfusion complications utilizing washed PRBC. Packed red blood cells (PRBC) will be washed at the blood bank to obtain MP depleted PRBC (PRBC-MP). A total of 500 patients undergoing CABG will be initially randomized to 2 groups: one to receive PRBC-MP, and the other conventional PRBC (PRBC+MP). Using a panel of lab tests/biomarkers selected for high sensitivity the investigators will compare the 2 groups with respect to subclinical physiologic host responses including (i) endothelial disturbances, (ii) inflammatory, and (iii) procoagulant responses. In addition, clinically evident transfusion complications and short term (<=30 days) surgical complications will be assessed and compared. Patients who are randomized but end up not requiring transfusion at surgery will serve as controls. Laboratory and clinical results will also be evaluated to elucidate which tests are significantly associated with clinically adverse effects.

SIGNIFICANCE. This study will shed new light on the biochemical and clinical effects of transfusion of MP. The findings of this investigation could significantly improve transfusion practice and safety.

DETAILED DESCRIPTION:
1. Study Design.

   1.1. Patient population. More than 500 coronary artery bypass surgeries (CABG) are performed annually at Jackson Memorial Hospital (JMH), the main teaching hospital of the U of M School of Medicine. The study coordinator works in close collaboration with Dr. Ricci, Co-Investigator. Dr. Ricci, working with other cardiac surgeons in his division, will screen all patients scheduled for CABG, and those who satisfy the eligibility criteria listed below will be invited to participate. Over a period of 37 months (between study months 4 and 41) 500 patients will be recruited and initially randomized to 2 groups: one (n=250) to receive conventional PRBC (unwashed PRBC) and the other (n=250) PRBC depleted of MP (washed PRBC). Approximately 50% of CABG will require PRBC transfusion during surgery and approximately 25% after surgery.

   The patient population can be further classified into the following subgroups: subgroup 1 (n=100), surgery transfusion with PRBC; subgroup 2 (n =100), surgery transfusion with washed PRBC; subgroup 3 (n =200), without any transfusion; subgroup 1a (n =25), surgery and post-surgery transfusion with PRBC ; subgroup 1b (n =25), no transfusion during surgery but post-surgery transfusion with PRBC; subgroup 2a (n =25), surgery and post surgery transfusion with washed PRBC; group 2b (n =25), no transfusion during surgery but post-surgery transfusion with washed PRBC.

   The comparison of major interest for this study is that of Subgroup 1 vs. 2, with approximately 100 patients each. -- Those not requiring transfusion (Subgroups 3, n ≈ 200) will serve as a "pure comparison" group. The remaining patients are those who require post surgery transfusion(s). The characteristics of patients in groups 1a, 1b, 2a, and 2b and their outcomes will be ascertained and they will be included in ancillary analyses. It is anticipated that only a small proportion of patients will require more than one post-surgery transfusion. Data pertaining to 2nd, 3rd, etc post-surgical transfusions will be collected and used for descriptive purposes and ancillary statistical analyses.

   1.2. Protocol on Transfusion Algorithm for the Washed PRBC Group.

   General Considerations

   Potential study participants will be screened and those satisfying the exclusion criteria, including patients with known platelet dysfunction or coagulopathy, will not be eligible for the trial. Once informed consent is signed, eligible candidates will be randomized to either of two approved transfusion practices: normal PRBC's or washed PRBC's.

   For patients randomized to the normal PRBC group, the usual blood bank procedures for transfusion will be followed during the pre-, intra-, and post-operative periods.

   For patients randomized to the washed PRBC group, the following general rules will be in place:

   Rule 1: PRBC's will be washed prior to surgery to avoid any delay in transfusion.

   Rule 2: The Blood Bank must be notified minimum 1 hour prior to transfusion, if more washed PRBC's are needed during or after surgery.

   Rule 3: Safety will never be compromised and the standard of care as applicable to blood transfusion requirements in coronary artery surgery patients will be preserved. In emergency situations, normal PRBC's will be transfused, if there is not enough time for PRBC washing.

   1.3. Blood sampling.

   Blood samples (in two tubes of citrated Vacutainers) will be obtained in all patients prior to induction of anesthesia, 1 hour after completion of surgery, and 1 and 7 days after surgery. Blood samples will be coded as follows:

   • BSa1, sample taken at induction of anesthesia • BSa2 1 hr post surgery • BSa3 at 1 day post-surgery • BSa4 at 7 days post surgery •

   Residual samples of every PRBC bag transfused, including that remaining in the tubing, will be obtained for MP profiling.
2. Main objectives of clinical study.

   The study is not designed to study major transfusion complications which are rare. The studies on biochemical physiologic host responses to the two types of PRBC are our main interest. They will be assessed by the sensitive assays previously described. Among patients showing abnormal test results, only a small fraction are expected to manifest clinically evident complications. The main objective of the clinical study is to asses these responses and compare the above described subgroups 1, 2 and 3 with respect to:

   2.1.Subclinical physiologic host responses including endothelial disturbance, procoagulant and proinflammatory responses, and oxidative stress;

   2.2. Minor or subtle post-transfusion reactions such as alteration of vital signs, cardiac disturbances, respiratory disturbances, O2 saturation; and in addition, short-term (<30 days) complications of cardiac surgery.

   2.3. A third aim is to assess correlation between laboratory biomarkers and clinical outcomes (minor transfusion reactions, short-term surgical outcomes), to gain insight into the mechanisms underlying adverse effects of transfusion and surgical complications. This will generate useful data on which tests or combination of tests best predict risk of complications of transfusion and surgery, regardless of whether they are found to be attributable to RMP or not.

   2.4. A fourth aim is to assess the mortality rate one year after surgery. This will be done by telephone, e-mail, or regular mail contact with the patients or their next of kin.
3. Patient recruitment; Randomization; pre-operative and perioperative care.

   3.1. Preoperative evaluation recruitment of patients. As normal part of preoperative evaluation, all cardiac surgery patients undergo complete medical history and physical examination, routine laboratory tests prior to a surgical procedure (including CBC, platelet count, chemistry, blood coagulation, lipid profiles, CRP, blood group), and cardiac evaluation including 2-D echocardiography and cardiac catheterization.

   All patients scheduled for CABG at JMH will be screened for eligibility. Medical records of all patients will be reviewed, and the following preoperative information will be evaluated and entered in the study data base: (1) Demographic and other characteristics including age, sex, race, blood type, body surface area (m2); (2) cardiac information: NYHA class I-IV, EKG, echocardiogram with ejection fraction; (3) preexisting medical conditions: hypertension, diabetes, chronic obstructive pulmonary disease, renal function, liver function, prior history of MI, stroke, peripheral vascular disease, thrombosis.

   Patients who satisfy the eligibility criteria listed below will be invited to participate in the study. The study coordinator will assist the Co-I with the entire process of recruitment and follow-up study. Prior to study enrollment, written informed consent will be obtained according to UM-IRB guidelines.

   3.2. Randomization. Once informed consent is signed, participants will be initially randomized to receive either packed red blood cells (PRBC) or washed packed cells (WPRBC). The randomization schedule will be prepared by Dr. Gomez using a block randomization scheme with varying block size. Copy of the randomization schedule will be provided to the study coordinator and the blood bank.

   Dynamic randomization scheme:

   To prevent potential imbalance between the two main groups due to the effect of some patients not requiring transfusion, a dynamic randomization scheme has been designed. Briefly, the randomization schedule will be designed to assign prospective patients sequentially to receive either washed or unwashed packed cells (PC). However, if any patient does not require a transfusion during surgery, this patient will be reassigned to Group 3 (non-transfusion) and will simply be skipped in the queue, and the next patient will be assigned to that position in the queue (since that position was not used due to no transfusion).
4. Laboratory assessments.

Overview. Subclinical physiologic responses (biomarkers) following transfusions will be assessed by laboratory studies. Broadly, the focus of interest is on sensitive markers of endothelial disturbance, procoagulant, proinflammatory, vasoactive and oxidative stress.

4.1. Routine blood tests will include CBC, platelets, reticulocyte counts, blood chemistry, C reactive protein (CRP), lipid profiles, DIC screen and tests for hemolysis.

4..2. Plasma MP. Total MP is measured by FITC-labeled lectin, Ulex; RMP by GlyPhA; PMP by CD41 and CD42+/CD31+; others as noted below.

4.3. Endothelial disturbance. (See Table C.1). Performed by assay of endothelial MP (EMP) using markers CD62E or CD31+/CD42- and EMP conjugates.

4.4. Procoagulant activities: All of the following reflect aspects of procoagulant activity: platelet activation marker CD62P; platelet MP (PMP) by CD42; total MP which are AnV+; total MP which are TF+; and MP-mediated thrombin generation (MP-TGA); Thrombin-antithrombin complex (TAT complexes).

4.5. Inflammatory markers. The following were selected as most informative. (i) Leukocyte MP (LMP) by flow cytometry: LMP are accepted by many investigators to reflect leukocyte activation, i.e., as inflammatory marker.

(ii) CD11b expression on leukocyte subsets. Widely accepted as a sensitive marker of leukocyte activation and inflammation. It is a simple and sensitive assay.

(iii) Platelet-leukocyte and EMP-leukocyte complexes are increasingly used as sensitive markers of inflammation.

(iv) Complement (C) activation. Detection of C components on MP by flow cytometry. Fragment C1q and C3 are measured on MP by flow cytometry. MP-associated IgG/IgM are of related interest and are measured in the PI's lab by FITC-goat anti-human Ab.

(v) Leukocyte nitric oxide (NO): Leukocyte NO is considered a marker of inflammation but also responds to oxidative state. In addition, it may reflect vascular tone since it is loosely coupled to plasma NO levels.

4.6. Other Biomarkers. (i). CD40L in plasma and MP-bound. CD40L, a marker both of inflammation and thrombosis, will be assayed by ELISA (Bender Med Systems).

(ii) Oxidative stress: ELISA kits which simplify the assay have become available at a reasonable cost. We have selected the kit from Assay Designs EIA because of good sensitivity (35 picrograms/mL).

(iii) Acetylcholinesterase (AChE) activity in plasma and MP.

4.7. Assay of MP from aliquots of PRBC transfused to patients. As stated earlier, residual blood from each PRBC bag transfused to patients will be obtained and analyzed for MP properties, e.g. total MP, RMP, contaminating MP (PMP, LMP, EMP), procoagulant activity, CD40L. This will enable verification of depletion of MP in washed PRBC's and assessment of any unusual properties that might be associated with adverse effects that may occur in the recipient.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring coronary artery bypass (CABG) surgery will be enrolled into the study if they: (1) are willing and able to give informed consent and to adhere to study follow up requirements; and (2) do not satisfy any of the exclusion criteria

Exclusion Criteria:

* Patients will be ineligible for the study if they (1) are unable or unwilling to give informed consent; (2) are unable or unwilling to follow the study protocol; (3) are less than 21 years of age; (4) require emergency procedures; (5) require cardiopulmonary bypass (pump) during the operation; (6) require other surgical procedures in addition to coronary artery bypass; (7) have a proven coagulation or platelet disorder; (8) are unwilling to receive blood transfusions; (9) are pregnant; or (10) have cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2010-07; Primary Completion 2014-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wenche Jy, PhD, Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States

REFERENCES:
- [Background] Horstman LL, Ahn YS. Platelet microparticles: a wide-angle perspective. Crit Rev Oncol Hematol. 1999 Apr;30(2):111-42. doi: 10.1016/s1040-8428(98)00044-4. No abstract available. PMID 10439058
- [Background] Horstman LL, Jy W, Jimenez JJ, Ahn YS. Endothelial microparticles as markers of endothelial dysfunction. Front Biosci. 2004 May 1;9:1118-35. doi: 10.2741/1270. PMID 14977533
- [Background] Koch CG, Li L, Sessler DI, Figueroa P, Hoeltge GA, Mihaljevic T, Blackstone EH. Duration of red-cell storage and complications after cardiac surgery. N Engl J Med. 2008 Mar 20;358(12):1229-39. doi: 10.1056/NEJMoa070403. PMID 18354101
- [Background] Piccin A, Murphy WG, Smith OP. Circulating microparticles: pathophysiology and clinical implications. Blood Rev. 2007 May;21(3):157-71. doi: 10.1016/j.blre.2006.09.001. Epub 2006 Nov 22. PMID 17118501
- [Background] Biro E, Nieuwland R, Tak PP, Pronk LM, Schaap MC, Sturk A, Hack CE. Activated complement components and complement activator molecules on the surface of cell-derived microparticles in patients with rheumatoid arthritis and healthy individuals. Ann Rheum Dis. 2007 Aug;66(8):1085-92. doi: 10.1136/ard.2006.061309. Epub 2007 Jan 29. PMID 17261534
- [Background] van den Goor JM, Nieuwland R, van Oeveren W, Rutten PM, Tijssen JG, Hau CM, Sturk A, Eijsman L, de Mol BA. Cell Saver device efficiently removes cell-derived microparticles during cardiac surgery. J Thorac Cardiovasc Surg. 2007 Sep;134(3):798-9. doi: 10.1016/j.jtcvs.2007.02.042. No abstract available. PMID 17723839
- [Derived] Jy W, Gomez-Marin O, Salerno TA, Panos AL, Williams D, Horstman LL, Ahn YS. Presurgical levels of circulating cell-derived microparticles discriminate between patients with and without transfusion in coronary artery bypass graft surgery. J Thorac Cardiovasc Surg. 2015 Jan;149(1):305-11. doi: 10.1016/j.jtcvs.2014.10.042. Epub 2014 Oct 14. PMID 25524686

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transfusion With Washed RBC | Transfusion With Unwashed RBC
Started | 73 | 104
Completed | 41 | 59
Not Completed | 32 | 45
Not completed — Adverse Event | 1 | 1
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 5
Not completed — Physician Decision | 29 | 35
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Hold by DSMB | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transfusion With Washed RBC | Transfusion With Unwashed RBC | Total
Number analyzed (Participants) | 41 | 59 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 30 | 54
  >=65 years | 17 | 29 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (7.1) | 63.9 (11.1) | 63.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 21 | 31
  Male | 31 | 38 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 33 | 60
  Not Hispanic or Latino | 14 | 26 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 14 | 24
  White | 31 | 43 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 59 | 100
CD41+ platelet microparticles [Mean (Standard Deviation); unit: counts / uL] — Cd41+ platelet microparticles is a specific biomarker for platelet activation
  counts / uL | 11858 (10066) | 12118 (10517) | 12009 (10279)
CD235a+ red cell microparticles [Mean (Standard Deviation); unit: counts / uL] — Cd235a+ red cell microparticles are a specific marker for red cell storage lesions. They may reflect the conditions of transfused RBC in circulation.
  counts / uL | 2017 (2414) | 1862 (1719) | 1927 (2029)
CD62E+ endothelial microparticles [Mean (Standard Deviation); unit: counts / uL] — CD62E+ endothelial microparticles are a specific marker for endothelial activation and apoptosis.
  counts / uL | 297 (430) | 296 (446) | 296 (435)
Annexin V+ microparticles [Mean (Standard Deviation); unit: counts / uL] — Annexin V+ microparticles are a marker for non-specific cell activation and apoptosis.
  counts / uL | 9171 (10710) | 6637 (6518) | 7697 (8568)

OUTCOME MEASURES:

1. Primary Outcome: In Hospital Mortality
Description: The number of participants who expired during hospital stay after CABG surgery
Time Frame: Within 30 days after CABG surgery
Measure: Number; unit: participants
Groups:
- Transfusion With Washed RBC: Subjects assigned to this arm were transfused with washed RBC
  Washed RBC: There is no pre-set dosage, frequency, or duration for transfusion with washed RBC. It all depends on the conditions of the patient during and after surgery. As circumstances arise, the physician will request needed washed RBC for the subject.
- Transfusion With Unwashed RBC: Subjects assigned to this arm were transfused with unwashed RBC
  Unwashed RBC: There is no pre-set dosage, frequency, or duration for transfusion with unwashed RBC. It all depends on the conditions of the patient during and after surgery. As circumstances arise, the physician will request needed unwashed RBC for the subject.
Arm/Group | Transfusion With Washed RBC | Transfusion With Unwashed RBC
Number analyzed (Participants) | 41 | 59
participants | 0 | 4
Statistical Analysis 1: Comparison: Transfusion With Washed RBC vs Transfusion With Unwashed RBC; Test type: Superiority or Other; p = 0.142, Fisher Exact

2. Primary Outcome: One-year Mortality
Description: Number participants who expired within one year after CABG surgery
Time Frame: Within one year after CABG surgery
Population: During the 12 months after hospital discharge, one participant in the group of transfusion with washed RBC and 3 participants in the group of transfusion with unwashed RBC were lost to follow up.
Measure: Number; unit: participants
Groups:
- Transfusion With Washed RBC: Subjects assigned to this arm were transfused with washed RBC
  Washed RBC: There is no pre-set dosage, frequency,or duration for transfusion with washed RBC. It all depends on the conditions of the patient during and after surgery. As circumstances arise, the physician will request needed washed RBC for the subject.
Arm/Group | Transfusion With Washed RBC | Transfusion With Unwashed RBC
Number analyzed (Participants) | 40 | 56
participants | 0 | 7
Statistical Analysis 1: Comparison: Transfusion With Washed RBC vs Transfusion With Unwashed RBC; Test type: Superiority or Other; p = 0.0391, Fisher Exact

3. Primary Outcome: Occurrence of at Least One Serious Adverse Event (SAE)
Description: Comparison of the two groups with respect to occurrence or not of at least one SAE including sepsis, respiratory failure, multi-organ failure, anaphylactic shock, transfusion-related acute lung injury, MI, stroke, cardiac arrest.
Time Frame: within 30 days after CABG surgery
Measure: Number; unit: participants
Arm/Group | Transfusion With Washed RBC | Transfusion With Unwashed RBC
Number analyzed (Participants) | 41 | 59
participants | 7 | 6
Statistical Analysis 1: Comparison: Transfusion With Washed RBC vs Transfusion With Unwashed RBC; Test type: Superiority or Other; p = 0.372, Fisher Exact

4. Primary Outcome: Difference in Levels of Circulating CD41+ Platelet-derived Microparticles 1 Hour Post-surgery
Description: Difference in levels of circulating CD41+ platelet microparticles between at pre-surgery and at 1hour post-surgery, i.e. level at 1hour post-surgery - level at pre-surgery
Time Frame: interval between presurgery and 1 hour post-surgery
Population: There were 2 participants' blood samples were not performed due to clotting or missing samples in the Group of "Transfusion with unwashed RBC". Therefore, the total number is 57 instead of 59 in that group.
Measure: Mean (Standard Deviation); unit: counts / uL
Arm/Group | Transfusion With Washed RBC | Transfusion With Unwashed RBC
Number analyzed (Participants) | 41 | 57
counts / uL | -1059 (9165) | 2034 (9077)
Statistical Analysis 1: Comparison: Transfusion With Washed RBC vs Transfusion With Unwashed RBC; Test type: Superiority or Other; p = 0.1007, t-test, 2 sided

5. Primary Outcome: Difference in Levels of Circulating Annexin V+ Microparticles 1 Hour Post- Surgery
Description: Difference in levels of circulating Annexin V+ microparticles between at pre-surgery and 1 hour post-surgery, i.e. level of Annexin V+ microparticles at 1 hour post-surgery - level of Annexin V+ microparticles at pre-surgery
Time Frame: Interval between pre-surgery and 1 hour post-surgery
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: counts / uL
Arm/Group | Transfusion With Washed RBC | Transfusion With Unwashed RBC
Number analyzed (Participants) | 40 | 57
counts / uL | -3589 (10940) | -680 (6022)
Statistical Analysis 1: Comparison: Transfusion With Washed RBC vs Transfusion With Unwashed RBC; Test type: Superiority or Other; p = 0.0964, t-test, 2 sided

6. Primary Outcome: Difference in Levels of Circulating CD62E+ Endothelial Microparticles 1 Hour Post-surgery
Description: Difference in levels of circulating CD62E+ endothelial microparticles between 1 hour post-surgery and at pre-surgery, i.e. level at 1 hour post-surgery - level at pre-surgery
Time Frame: Interval between pre-surgery and 1 hour post-surgery
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: counts / uL
Arm/Group | Transfusion With Washed RBC | Transfusion With Unwashed RBC
Number analyzed (Participants) | 41 | 57
counts / uL | 36.4 (176.5) | 2.0 (59.1)
Statistical Analysis 1: Comparison: Transfusion With Washed RBC vs Transfusion With Unwashed RBC; Test type: Superiority or Other; p = 0.1739, t-test, 2 sided

7. Primary Outcome: Difference in Levels of Circulating CD235a+ Red Cell Microparticles 1 Hour Post-surgery
Description: Difference in levels of circulating CD235a+ red cell microparticles between at 1 hour post-surgery and at pre-surgery, i.e. levels at 1 hour post-surgery - level at pre-surgery
Time Frame: Interval between pre-surgery and 1 hour post-surgery
Measure: Mean (Standard Deviation); unit: counts / uL
Arm/Group | Transfusion With Washed RBC | Transfusion With Unwashed RBC
Number analyzed (Participants) | 41 | 57
counts / uL | -344 (2576) | -208 (1070)
Statistical Analysis 1: Comparison: Transfusion With Washed RBC vs Transfusion With Unwashed RBC; Test type: Superiority or Other; p = 0.7205, t-test, 1 sided

8. Secondary Outcome: Each Participant's Number of Non-serious Adverse Events
Description: All clinical non-serious adverse events reported in the clinical chart were recorded in the study's data files. This type of events, defined as Non-Serious Adverse Events or just Adverse Events (AEs) were categorized into 5 groups: (1) Cardiovascular / respiratory; (2) renal; (3) neurologic (CNS); (4) infections; and (5) other. For each participant, the outcome measure was defined as the number of AE's he or she experienced during his/her hospital stay.
Time Frame: Within 30 days after CABG surgery
Measure: Mean (Standard Deviation); unit: Adverse events
Arm/Group | Transfusion With Washed RBC | Transfusion With Unwashed RBC
Number analyzed (Participants) | 41 | 59
Adverse events | 1.5 (1.1) | 2.4 (2.2)
Statistical Analysis 1: Comparison: Transfusion With Washed RBC vs Transfusion With Unwashed RBC; Test type: Superiority or Other; p = 0.0176, t-test, 2 sided; Negative Binomial = 1.64, 95% CI 2-sided [1.06 to 2.55] — Using Negative Binomial Regression the following ratio and corresponding 95% CI were obtained: (# of AE's, Unwashed Group / (# of AE's, Washed Group) = 1.64 95% C.I. = [1.06 - 2.55]

ADVERSE EVENTS:
Time Frame: Within 30 days after CABG surgery
Arm/Group | Transfusion With Washed RBC | Transfusion With Unwashed RBC
Serious Adverse Events (participants affected / at risk) | 7/41 | 6/59
Other Adverse Events (participants affected / at risk) | 21/41 | 44/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transfusion With Washed RBC (N=41) | Transfusion With Unwashed RBC (N=59)
MI (Cardiac disorders) | 5 (5) | 4 (4)
Renal Failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transfusion With Washed RBC (N=41) | Transfusion With Unwashed RBC (N=59)
Neurologic AE (Nervous system disorders) | 7 (7) | 10 (10)
CVD (Vascular disorders) | 16 (16) | 31 (31)
Infection (Infections and infestations) | 3 (3) | 4 (4)
Renal (Renal and urinary disorders) | 1 (1) | 7 (7)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 18 (18)
Thrombosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Fever (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
A major limitation of the present study is its small sample size and its restriction to CABG surgery. Larger-scale controlled studies comparing transfusion with washed vs. unwashed PCs are warranted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No